CLINICAL TRIAL: NCT03729349
Title: Golimumab for Adherence in Rheumatoid Arthritis
Acronym: GO FAR
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108555; CNTO148ARA4010 (Other: Janssen Inc.)
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Diagnosis of Rheumatoid Arthritis: Participants will not receive any intervention as a part of this study. All Rheumatoid Arthritis (RA) participants treated with golimumab in a clinical practice setting will be observed.
  Interventions: Biological: Golimumab

INTERVENTIONS:
Biological: Golimumab — Participants will receive golimumab as a part of clinical practice.
  Other Names: SIMPONI ™

SUMMARY:
The purpose of this study is to determine if non-adherence to Rheumatoid Arthritis (RA) drugs in participants treated with biologic disease modifying anti-rheumatic drugs (DMARDs) is associated with a greater incidence of disease in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of rheumatoid arthritis
* About to initiate therapy with golimumab
* Must sign a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Diagnosis of Axial Spondyloarthritis, Ankylosing Spondylitis or Psoriatic Arthritis
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the start of the study or the first data collection time point
* Currently enrolled in an investigational study
* Currently enrolled in an observational study sponsored or managed by a Janssen company

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Rheumatoid Arthritis (RA) participants treated with golimumab in a clinical practice setting will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Impact of Adherence on Flares as Assessed by Rheumatoid Arthritis Flare Questionnaire (RA-FQ) Score at 6 Month | 6 Month
  Impact of adherence on flares will be assessed by RA-FQ score or the answer to question 7 of the RA-FQ (Are you having a flare?) at 6 month in participants categorized as "low predicted compliance" vs "high predicted compliance". RA-FQ is 10 point scale for questions 1 to 5, with score range from 0 to 10, where higher score indicates worse outcome and having option 'Yes' and 'No' for question 6 and 7. The RA-FQ total score is calculated as the sum of responses for items 1-5 (maximum 50). Higher score indicates worst outcome.
Impact of Adherence on Flares as Assessed by RA-FQ Score at 12 Month | 12 Month
  Impact of adherence on flares will be assessed by RA-FQ score or the answer to question 7 of the RA-FQ (Are you having a flare?) at 12 month in participants categorized as "low predicted compliance" vs "high predicted compliance". RA-FQ is 10 point scale for questions 1 to 5, with score range from 0 to 10, where higher score indicates worse outcome and having option 'Yes' and 'No' for question 6 and 7. The RA-FQ total score is calculated as the sum of responses for items 1-5 (maximum 50). Higher score indicates worst outcome.

SECONDARY OUTCOMES:
Percentage of Adherent Participants at 6 and 12 Months | Months 6 and 12
  Percentage of adherent participants at 6 and 12 Months will be assessed.
Number of Participants with Corticosteroid Use | Months 6 and 12
  Number of participants with corticosteroid use will be assessed among participants categorized as "low predicted compliance" vs "high predicted compliance" at 6 and 12 months.
Predicting Factors for Adherence | Months 6 and 12
  Independent predictors of "predicted compliance" will be assessed with univariate and multivariate Cox regression analysis.
Number of Participants with any Adverse Events (AEs), Serious Adverse Events (SAEs) or Discontinuation of Golimumab | Months 6 and 12
  Number of participants with any AEs, SAEs or discontinuation of golimumab will be assessed among participants categorized as "low predicted compliance" vs "high predicted compliance" at 6 and 12 months and include any such event up to the previous study visit.
Percentage of Participants with Response to Patient Support Program Question | Months 6 and 12
  Percentage of participants with response to Patient Support Program Question (Yes/No) will be assessed among participants categorized as "low predicted compliance" vs "high predicted compliance" at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (32):
- Canada (32):
  - Peak Medical Specialty Centre, Calgary, Alberta
  - Jacqueline C Stewart Medical Inc., Penticton, British Columbia
  - Dr. Milton F Baker Inc., Victoria, British Columbia
  - Fredericton Medical Clinic, Fredericton, New Brunswick
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - St Clare's Hospital, St. John's, Newfoundland and Labrador
  - Private Practice - Dr. Diane Wilson, Lunenburg, Nova Scotia
  - The Waterside Clinic, Barrie, Ontario
  - Dr. Sankalp V. Bhavsar Medicine Professional Corporation, Burlington, Ontario
  - Private Practice - Dr. Pauline Boulos, Dundas, Ontario
  - Dr. Sangeetha Thiviyarajah Medicine Professional Corporation, Etobicoke, Ontario
  - Samuel Silverberg Medicine Professional Corporation, Etobicoke, Ontario
  - Adachi Medicine Professional Corporation, Hamilton, Ontario
  - Manisha Mulgund Medicine Professional Corporation, Hamilton, Ontario
  - K-W Musculoskeletal Research Inc, Kitchener, Ontario
  - Markham Rheumatology Hub, Markham, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario
  - Dr. Rajwinder S Dhillon Medicine Professional Corporation, Niagara Falls, Ontario
  - Makhzoum Medicine Professional Coporation, Oakville, Ontario
  - Dr. S. Gill Medicine Professional Corporation, Oakville, Ontario
  - Dr. Abraham Chaiton Medicine Professional Corporation, Toronto, Ontario
  - Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Arthur Karasik Medicine Professional Corporation, Toronto, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Clinique de Rhumatologie de Montreal, Montreal, Quebec
  - Private Practice Dr Louis Bessette, Québec, Quebec
  - Centre de sante et services sociaux (CSSS) de Rimouski-Neigette - Hopital regional - Rimouski, Rimouski, Quebec
  - CIUSSS de L Estrie CHUS, Sherbrooke, Quebec
  - Clinique Jacques Cartier- Rheumatology Division - Université de Sherbrooke, Sherbrooke, Quebec
  - Centre de Recherche Musculo Squelettique, Trois-Rivières, Quebec
  - Community Rheumatology Care, Saskatoon, Saskatchewan
  - Rheumatology Associates of Saskatoon, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Bessette L, Boulos P, Arendse R, Rahman P, Aseer S, Ruban T, Rachich M, Nantel F, Calce A, Asin-Milan O, Haaland D. Impact of Adherence to Golimumab on Disease Flares in Rheumatoid Arthritis: Results from a Canadian Observational Study. Patient Prefer Adherence. 2025 Jun 25;19:1843-1853. doi: 10.2147/PPA.S516794. eCollection 2025. PMID 40585577